CLINICAL TRIAL: NCT03765424
Title: Evaluation of Ultrasound and PET/CT in the Diagnosis and Monitoring of Giant Cell Arteritis
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: The Danish Rheumatism Association (Other); Hartmann Fonden (Other); AP Moeller Foundation (Other); Aase and Ejnar Danielsens Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ULvsPET GCA cohort
Record Dates: First submitted 2018-11-28; First posted 2018-12-05 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2018-11

CONDITIONS: Giant Cell Arteritis; Vasculitis
MeSH Terms: conditions — Giant Cell Arteritis; Vasculitis | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Full blood EDTA plasma Lithium-heparin plasma serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GCA cases: GCA cases were patients with a clinical diagnosis of GCA based on a rheumatologists evaluation of history taking, physical examination, laboratory screening and initial PET report (reporting potential large vessel inflammation but not considering cranial artery inflammation).
  GCA was considered large vessel (LV) and/or cranial (c) GCA cases:
  LV-GCA cases were patients with a clinical diagnosis of GCA and verified LV inflammation by 18F-FDG PET/CT with or without concomitant c-GCA.
  C-GCA cases, for the exploratory analysis of the performance of US and PET in c-GCA, were patients with a clinical diagnosis of GCA fulfilling the 1990 American College of Rheumatology (ACR) criteria, with or without concomitant LV-GCA.
  Interventions: Diagnostic Test: Ultrasound
- controls: Controls were GCA suspected patients in whom GCA diagnosis was dismissed.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Ultraosund of temporal, carotid and axillary arteries

SUMMARY:
The aim of this project is to prospectively evaluate the diagnostic accuracy of different imaging tools in specific giant cell arteritis disease subsets before and after treatment initiation. Diagnostic tools with high sensitivity and specificity are a prerequisite for optimal treatment of GCA patients.

Specifically, the diagnostic accuracy of ultrasound (US) as compared to 18F-FDG PET/CT in new-onset, treatment naïve large vessel(LV)-GCA patients is investigated. Furthermore, long-term follow up including US, 18F-FDG PET/CT and cross sectional imaging is performed to explore the potential of imaging as monitoring and prognostic tools.

In this observational cohort, the diagnostic accuracy of 18F-FDG PET/CT after three and ten days of glucocorticoid treatment in the subset of LV-GCA patients and the diagnostic accuracy of 18F-FDG PET/CT in cranial artery inflammation in new-onset, treatment naïve c-GCA patients as compared to a control group of patients with a previous diagnosis of malignant melanoma was also evaluated and is registered elsewhere (ClinicalTrials.gov Identifier: NCT03285945 and NCT03409913, respectively)

DETAILED DESCRIPTION:
The diagnosis of GCA is clinical and syndrome-based. Only few years ago, temporal artery biopsy (TAB) was the standard diagnostic tool to confirm diagnosis, although sensitivity is moderate[3,4] and its outcome seldom affects treatment management[5]. Today, the European League Against Rheumatism (EULAR) recommends diagnostic imaging in all patients suspected of GCA[6]. The imaging of choice is based on the suspected vessel involvement. In patients suspected of cranial GCA (c-GCA), vascular ultrasound (US) is the recommended first line imaging test, whereas Fluorine-18-fluorodeoxyglucose (18F-FDG) positron emissions tomography/computed tomography (PET/CT) is not recommended for the assessment of cranial arteries.

In patients suspected of large vessel involvement (LV-GCA), 18F-FDG PET/CT, US, magnetic resonance imaging (MRI) or CT can be used to confirm disease, but no specific priority of the imaging tests is given. US is an attractive first line imaging in LV-GCA suspected patients since it is increasingly used in the diagnosis of c-GCA, is readily available and cheap. 18F-FDG PET/CT is an appealing diagnostic tool in LV-GCA suspected patients, since it also evaluates malignancy and infection, differential diagnoses often considered in this disease subset. However, 18F-FDG PET/CT is often not readily available, is expensive and exposes patients to radiation. Moreover, its sensitivity seems to decrease with glucocorticoid (GC) treatment and the window of opportunity in which sensitivity is unaffected is unknown.

Relapse during glucocorticoid tapering is frequent in GCA. However, the evaluation of potential GCA disease activity relies on unspecific symptoms and inflammatory biomarkers. There is a significant overlap between symptoms of GCA disease activity and GC adverse effect and the same holds for symptoms and biomarkers of disease activity and infection, making the evaluation difficult. Accurate tools to support treatment decisions, avoid over-treatment without risk of GCA related complications are lacking.

The aim of this project is to prospectively evaluate the diagnostic accuracy of different imaging tools in specific giant cell arteritis disease subsets before and after treatment initiation. Diagnostic tools with high sensitivity and specificity are a prerequisite for optimal treatment of GCA patients.

Specifically, the diagnostic accuracy of ultrasound (US) as compared to 18F-FDG PET/CT in new-onset, treatment naïve large vessel(LV)-GCA patients is investigated. Furthermore, long-term follow up including US, 18F-FDG PET/CT and cross sectional imaging is performed to explore the potential of imaging as monitoring and prognostic tools.

In this observational cohort, the diagnostic accuracy of 18F-FDG PET/CT after three and ten days of glucocorticoid treatment in the subset of LV-GCA patients and the diagnostic accuracy of 18F-FDG PET/CT in cranial artery inflammation in new-onset, treatment naïve c-GCA patients as compared to a control group of patients with a previous diagnosis of malignant melanoma was also evaluated and is registered elsewhere (ClinicalTrials.gov Identifier: NCT03285945 and NCT03409913, respectively)

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 50 years
2. C-reactive protein (CRP)>15 mg/L or erythrocyte sedimentation rate (ESR)>40 mm/h
3. Either

   1. cranial symptoms such as new-onset headache or scalp tenderness, jaw or tongue claudication, visual disturbances
   2. new-onset limb claudication
   3. protracted constitutional symptoms, defined as weight loss>5 kilograms or fever>38 degrees Celcius for >3 weeks
   4. Bilateral shoulder pain and morning stiffness.

Exclusion Criteria:

1. oral glucocorticoid treatment within the past month;
2. subcutaneous, intramuscular, intra-articular or intravenous glucocorticoid within the past 2 months;
3. DMARD treatment or other immunosuppressive therapy within the past 3 months;
4. ongoing treatment with interleukin2;
5. previous diagnosis of GCA or polymyalgia rheumatica;
6. any disease potentially causing large vessel inflammation, that is autoimmune diseases; rheumatoid arthritis, Cogans syndrome, relapsing polychondritis, ankylosing spondylitis, systemic lupus erythematosus, Buerger's disease, Bechet's disease, inflammatory bowel disease, infections; syphilis, known active current or history of recurrent tuberculosis, hepatitis or HIV, or other large vessel disease; sarcoidosis, neurofibromatosis, congenital coarctation, Marfans syndrome, Ehlers-Danlos syndrome, retroperitoneal fibrosis.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the GCA suspect cohort, patients referred to Department of Rheumatology, Aarhus University Hospital due to suspicion of GCA are considered for inclusion. Patients in whom a 18F-FDG PET/CT is not performed by the time of referral and who presents with unequivocal cranial symptoms of GCA requiring acute initiation of GC treatment are not considered for inclusion.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of large vessel ultrasound with PET/CT as reference | Time of diagnosis/pre-treatment
  Large vessel ultrasound for LV-GCA diagnosis is considered positive in the presence of a halo in carotid and/or axillary arteries.

SECONDARY OUTCOMES:
Large vessel intima-media thickness (IMT) cut off for LV-GCA diagnosis with PET/CT as reference | Time of diagnosis/pre-treatment
  IMT measurement performed on the distal vessel wall in carotid and axillary arteries
Diagnostic accuracy vascular ultrasound (overall) | Time of diagnosis/pre-treatment
  Vascular ultrasound for GCA diagnosis is considered positive in the presence of a halo in temporal, carotid and/or axillary arteries.
Diagnostic accuracy of vascular ultrasound after treatment (day 3, 10 and week 8) | 3 days, 10 days and 8 weeks after initiated treatment
  Vascular ultrasound for GCA diagnosis is considered positive in the presence of a halo in temporal, carotid and/or axillary arteries.
Diagnostic accuracy of PET/CT of cranial arteries for c-GCA diagnosis (reference: American College of Rheumatology 1990 criteria) | Time of diagnosis/pre-treatment
  cranial artery (vertebral, maxillary and temporal) FDG uptake above surrounding tissue FDG uptake is considered consistent with vasculitis
Temporal artery biopsy | Time of diagnosis
  Temporal artery biopsy considered positive in the presence of an inflammatory infiltrate in any vessel wall layer
Halo sign for monitoring disease activity (week 8, 24 and 15 months) | week 8, 24 and 15 months after initiated treatment
  Presence or absence of halos on US
Composite halo score for monitoring disease activity (week 8, 24 and 15 months) | week 8, 24 and 15 months after initiated treatment
  Composite halo score
Intima media thickness for monitoring disease activity (week 8, 24 and 15 months) | week 8, 24 and 15 months after initiated treatment
  Maximum intima media thickness (IMT) measurement on US
PETVAS for monitoring disease activity (15 months) | 15 months after treatment is initiated
  Composite PET scores (e.g.PETVAS)
Semiquantitative FDG measure for monitoring disease activity (15 months) | 15 months after treatment is initiated
  Maximum semiquantitative FDG measures
FDG burden for monitoring disease activity (15 months) | 15 months after treatment is initiated
  Composite scores of FDG inflammatory burden (summarising FDG uptake in voxels of interest)
PETVAS for GCA prognosis (baseline) | 4-5 years after diagnosis
  PETVAS score (summarising graded (1-4) FDG uptake in arterial vessel segments)
Semiquantitative FDG measure for GCA prognosis (baseline) | 4-5 years after diagnosis
  Maximum semiquantitative FDG measures
FDG burden for GCA prognosis (baseline) | 4-5 years after diagnosis
  Composite scores of arterial FDG uptake (summarising FDG uptake in voxels of interest)
Aortic diameter 4-5 years after diagnosis | 4-5 years after diagnosis
  Aortic diameter on cross sectional imaging
Vessel wall thickening 4-5 years after diagnosis | 4-5 years after diagnosis
  Vessel wall thickening

OTHER OUTCOMES:
Patient global NRS | Baseline, day 10, week 8, 24 and 15 months
  Patients global experience of disease activity on a numerical range scale (0-10)
Physician NRS | Baseline, day 10, week 8, 24 and 15 months
  Physicians global judgement of disease activity on a numerical range scale (0-10)
CRP | Baseline, day 3 and 10, week 8, 24 and 15 months
  c-reactive protein (mg/l)
Physicians judgement of disease activity | Baseline, day 10, week 8, 24 and 15 months
  Overall judgement of disease activity (remission, possible activity not requiring treatment, activity/relapse)
Cumulated glucocorticoid dose | Baseline, day 10, week 8, 24 and 15 months
  Cumulated glucocorticoid dose (mg)
Glucocorticoid dose | Baseline, day 10, week 8, 24 and 15 months
  Glucocorticoid dose (mg)
Cardiovascular events | 4-5 years
  Cardiovascular events (number)

CONTACTS AND LOCATIONS:
Overall Officials: Berit Nielsen, MD, Principal Investigator — Department of Rheumatology

IPD SHARING:
Plan to Share IPD: No